CLINICAL TRIAL: NCT04134130
Title: Case Control Study Regarding the Role of Follicle Stimulating Hormone in Chemically Castrated Young Men
Brief Title: The Role of Follicle Stimulating Hormone in Advanced Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Swedish Cancer Foundation (Other); ALF Swedish Government Grant (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-01942
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer Recurrent
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Gonadotropins; testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: Randomized case control study: one arm with FSH treatment for 5 weeks and one arm without FSH.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GnRH antagonist + FSH + testosterone (Other): At the start of the study: 240 mg of the gonadotropin releasing hormone antagonist Degarelix (Ferring GmbH, Wittland, Kiel, Germany) + recombinant FSH (Gonal-f, Merck Serrono S.A. Aubonne, Schweiz), 300 IU every second day for 5 weeks.
  After 3 weeks: 1000 mg testosterone once.
  Interventions: Drug: Degarelix 120 MG [Firmagon]; Drug: Gonal F RFF Pen 900 UNT Per 1.5 ML Pen Injector; Drug: Testosterone Undecanoate
- GnRH antagonist + testosterone (Other): At the start of the study: 240 mg of the gonadotropin releasing hormone antagonist Degarelix (Ferring GmbH, Wittland, Kiel, Germany).
  After 3 weeks: 1000 mg testosterone (Nebido, Bayer AB, Solna, Sweden) once.
  Interventions: Drug: Degarelix 120 MG [Firmagon]; Drug: Testosterone Undecanoate

INTERVENTIONS:
Drug: Degarelix 120 MG [Firmagon] — Two doses of degarelix, 240 mg, subcutaneously once, at study start.
  Other Names: Firmagon
Drug: Gonal F RFF Pen 900 UNT Per 1.5 ML Pen Injector — Gonal-f 300 IU subcutaneously 3 times per week for 5 weeks.
  Other Names: Gonadotropin
  Arms: GnRH antagonist + FSH + testosterone
Drug: Testosterone Undecanoate — One dose 1000 mg testosterone once, after 3 weeks.
  Other Names: Nebido

SUMMARY:
In order to elucidate if FSH can have testosterone like effects, samples from young, non-smoking healthy volunteers, with normal body mass index, and with pharmacologically induced gonadotropin deficiency will be studied regarding their capacity to induce prostate specific antigen (PSA), which normally is regulated by testosterone.

DETAILED DESCRIPTION:
Normally, prostate specific antigen (PSA), which is a marker for prostate disease and progression, is exclusively produced in response to testosterone. In order to elucidate if follicle stimulating hormone (FSH) can have testosterone like effects, samples from n=30 non-smoking healthy volunteers, 20-30 years of age and with normal body mass index (20-25) with pharmacologically induced gonadotropin deficiency will be studied. The men are currently recruited and during 5 weeks undergoing:

1. Pharmacologically induced gonadotropin deficiency w 1-3;
2. FSH-treatment of 50% (group A), w 1-5;
3. Testosterone (T) treatment of all (group A and B) w 4-5;
4. End and follow up after 5 weeks.

A subcutaneous injection with the GnRH antagonist degarelix (240 mg¸ Ferring GmbH Wittland, Kiel, Germany) results in drop of both FSH and LH-induced testosterone. Half of the men will get recombinant FSH (300 IU; Gonal-f, Merck Serrono S.A. Aubonne, Schweiz) back, whereas 50% will not. Three weeks thereafter, the full spectrum of FSH dependent changes occur and are reflected in blood. From this occasion testosterone (Nebido, Ferring GmbH Wittland, Kiel, Germany) will be given to all participants to diminish the side-effects of the castration. Blood samples are collected at start, after 3 wks and after 5 wks. At that point also a follow up is undertaken. This experimental design will provide samples from each individual during normal conditions, during castration, and after a standardised dose of FSH.

ELIGIBILITY:
Inclusion Criteria: Healthy, non-smoking, body mass index 20-25, Exclusion Criteria: Medication or drug abuse

-

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
PSA-concentration | 5 weeks
  Prostate marker

SECONDARY OUTCOMES:
FSH dependent proteins | 5 weeks
  Proteins identified by spectrophotometry

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lundberg Giwercman, Professor, Principal Investigator — Lund University, dept Translational medicine
Locations (1):
- Reproductive Medicine Center, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No